CLINICAL TRIAL: NCT00803309
Title: Optimization of Treatment for Patients With Chronic Hepatitis C Infected With HCV-genotype 2 or 3: 12 vs. 24 Weeks of Treatment Extension for Patients Without Rapid Virological Response
Brief Title: Study to Assess the Efficacy of 12 Versus 24 Weeks of Extended Treatment in HCV-Genotype 2/3 Patients
Acronym: OPTEX2/3
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: At the end of the planned recruitment period the expected number of subjects could not be included in the trial.
Sponsor: HepNet Study House, German Liverfoundation (Network)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05498
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic HCV-genotype 2/3; Efficacy of treatment extension; PegIntron; pegylated interferon alpha-2b; Rebetol; ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): PegIntron® 1.5 µg/kg once weekly (QW) subcutaneous (sc) plus Rebetol® 800-1400 mg per os divided in 2 daily doses for additional 24 weeks beyond standard treatment with 24 weeks follow-up
  Interventions: Drug: pegylated interferon alpha-2b; Drug: Ribavirin
- B (Active Comparator): PegIntron® 1.5 µg/kg QW sc plus Rebetol® 800-1400 mg per os divided in 2 daily doses for additional 12 weeks beyond standard treatment with 24 weeks follow-up
  Interventions: Drug: pegylated Interferon alpha-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha-2b — 1.5 µg/kg once weekly, syringe, 24 weeks
  Other Names: PegIntron
  Arms: A
Drug: Ribavirin — 800-1400 mg per os, daily, tablets, 24 weeks
  Other Names: Rebetol
  Arms: A
Drug: pegylated Interferon alpha-2b — 1.5 µg/kg once weekly, syringe, 12 weeks
  Other Names: PegIntron
  Arms: B
Drug: Ribavirin — 800-1400 mg per os, daily, tablets, 12 weeks
  Other Names: Rebetol
  Arms: B

SUMMARY:
In this study we intend to treat patients with chronic hepatitis C of genotype 2 or 3 having characteristics associated with poor treatment response for additional 12 or 24 weeks beyond the standard treatment of PEG-IFN alpha-2b plus ribavirin.

The objective of this study is to compare the efficacy of a treatment extension of 12 versus 24 weeks in patients with HCV-genotypes 2 and 3 who are treated with 1.5 µg/kg PEG-IFN alpha-2b and 800-1400 mg ribavirin (standard dose) for 24 weeks (standard duration) and who are not HCV-RNA negative (< 15 IU/ml) after 4 weeks of standard treatment but HCV-RNA negative after 16-24 weeks of standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with HCV-genotype 2/3 chronic hepatitis C documented by detectable plasma HCV RNA (> 15 IU/mL) and positivity of anti-HCV antibodies
* Age ≥ 18 years
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Negative urine or blood pregnancy test (one of the both; for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug. Additionally, all fertile males and females must be using two forms of effective contraception during treatment and during the 7 months after treatment end. This includes using birth control pills (no interaction with investigational drugs), IUDs, condoms, diaphragms, or implants, being surgically sterilized, or being in a post-menopausal state. At least one contraception method must be of barrier method
* Ongoing treatment with 1.5 µg/kg Peg-Interferon alpha-2b (PegIntron®) and > 10.6 mg/kg ribavirin (Rebetol®)
* No rapid virological response (HCV-RNA positive after week 4 of the ongoing therapy)
* Willingness to give written informed consent and willingness to participate to and to comply with the study protocol

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Male partners of women who are pregnant
* Positive tests at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, HBeAg, anti-HIV, HIV-RNA
* History or other evidence of a medical condition associated with chronic liver disease other than HCV associated (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposures)
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Patients with liver cirrhosis with a lesion suspicious for hepatic malignancy on the screening
* Absolute neutrophil count (ANC) <750 cells/mm3 at screening
* Platelet count <50,000 cells/mm3 at screening
* Hb <10 g/dl at screening
* Dose modification of Peg-Interferon alpha-2b (PegIntron®) or ribavirin (Rebetol®) during the first 4 weeks of the ongoing therapy
* Interferon alpha or ribavirin therapy at any time point before the actual ongoing treatment
* Less than 80% adherence to treatment of the ongoing treatment until randomization (week 20-22 of ongoing treatment)
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression (ICD 10 codes F30-F33). Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time. Patients are excluded if any history of suicidal attempts is evident. If hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease are documented, psychiatric consultation is mandatory. Patients with a mild or moderate psychiatric disease (ICD 10 codes F32.0, F32.1, F33.0, F33.1) are only allowed to be included into the trial if a regular monitoring by a psychiatrist is performed during the trial
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis)
* History or any other evidence of autoimmune diseases
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of significant cardiac disease that could be worsened by acute anemia (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months prior to treatment with Peg-Interferon/ribavirin therapy, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina)
* Evidence of thyroid disease that is poorly controlled on prescribed medications
* Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration)
* History of major organ transplantation with an existing functional graft
* History or other evidence of severe illness, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Patients with evidence for tuberculosis
* Drug abuse within 6 months prior to the first dose of study drug and excessive alcohol consumption. Patients on methadone/polamidone/buprenorphine programs are not excluded
* Any investigational drug and/or participation in another clinical study prior 6 months to the actual ongoing antiviral treatment
* Limited contractual capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Reduction of Relapse rate (HCV-RNA positive in serum by a standard HCV-PCR with a detection limit of at least 15 IU/ml) 24 weeks after the end of treatment and thus improvement of sustained virological response rates (SVR) | 48 weeks (arm A) or 36 weeks (arm B)

SECONDARY OUTCOMES:
Virological response rates (HCV-RNA negative in serum by a standard HCV-PCR with a detection limit of at least 15 IU/ml) at the end of therapy | 24 weeks (arm A) or 12 weeks (arm B)
Biochemical responses as determined by ALT and AST levels at the end of treatment and at the end of follow up. | Arm A: 24 and 24 weeks, arm B: 12 and 24 weeks
Severity and frequency of adverse event | 48 weeks (arm A) or 36 weeks (arm B)
Analysis of quality of life | 48 weeks (arm A) or 36 weeks (arm B)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Manns, Prof. Dr., Study Director — Hannover Medical School
Locations (49):
- Germany (49):
  - Ärztehaus Leipziger Straße, Berlin
  - Medizinisches Infektiologiezentrum, Berlin
  - Praxis Dr. med. Naumann, Berlin
  - Hepatologische Schwerpunktpraxis im bng, Berlin
  - Charité Campus Virchow-Klinikum, Med. Klinik für Gastroenterologie und Hepatologie, Berlin
  - Praxis Dr. med. J. Gölz, Berlin
  - Praxis Meyer, Berlin
  - Friedrich-Wilhelms-Universität, Med. Klinik und Poliklinik I, Bonn
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Kreiskliniken Burghausen/Altötting, Med. Klinik II, Burghausen/Altötting
  - Hepatologische Schwerpunktpraxis im bng, Dortmund
  - Krankenhaus Dresden-Friedrichstadt, Dresden
  - Fachärztliche Gemeinschaftspraxis, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum der J.W. Goethe-Universität, Frankfurt
  - Vitanus GmbH, Frankfurt
  - Praxis Zentrum Gastroenterologie und Endokrinologie, Freiburg im Breisgau
  - Asklepios Klinik St. Georg, Institut für interdiziplinäre Infektiologie, Hamburg
  - IPM-Studycenter GmbH & Co. KG, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Innere Medizin, Hamburg
  - Universtätsklinikum Hamburg-Eppendorf;Innere Medizin, Hamburg
  - Praxis Dr. med. S. Holm, Hanover
  - Leberpraxis Hannover, Hanover
  - Medizinische Hochschule Hannover, Zentrum Innere Medizin, Hanover
  - Medizinische Fakultät der Universität Heidelberg, Innere Medizin IV, Heidelberg
  - Hepatologische Schwerpunktpraxis im bng, Herne
  - Universitätskliniken des Saarlandes, Innere Medizin II, Gastroenterologie, Homburg
  - Klinik für Innere Medizin der FSU, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Allgemeine Innere Medizin, Kiel
  - Gastroenterologische Gemeinschaftspraxis, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Gemeinschaftspraxis Dr.Simon, Leverkusen
  - Universitätklinikum Schleswig-Holstein, Campus Lübeck, Med. Klinik I, Lübeck
  - Otto-von-Guericke Universität Magdeburg, Magdeburg
  - Klinikum der Johannes Gutenberg Universität Med. Klinik, Mainz
  - Universitäts-Klinikum Mannheim, Med. Klinik II, Mannheim
  - Hepatologische Schwerpunktpraxis im bng, Minden
  - Klinikum Großhadern, Med. Klinik 2, München
  - Universitätsklinikum Münster, Med. Klinik und Poliklinik B, Münster
  - St.-Theresien-Krankenhaus, Nuremberg
  - St. Josef Hospital, Oberhausen
  - Hepatologische Schwerpunktpraxis im bng, Offenbach
  - St.-Josefs-Klinik, Med. Klinik, Offenburg
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Medizin I, Regensburg
  - Diakoniekrankenhaus, Med. Klinik II, Rotenburg (Wümme)
  - Praxis Dr. med. A. Trein, Stuttgart
  - Universitätsklinikum Tübingen Medizinische Klinik I, Tübingen
  - Universitätsklinikum Ulm, Abteilung für Innere Medizin I, Ulm
  - Med. Poliklinik der Universität Würzburg, Würzburg

REFERENCES:
- [Result] Heidrich B, Cordes HJ, Klinker H, Moller B, Naumann U, Rossle M, Kraus MR, Boker KH, Roggel C, Schuchmann M, Stoehr A, Trein A, Hardtke S, Gonnermann A, Koch A, Wedemeyer H, Manns MP, Cornberg M. Treatment Extension of Pegylated Interferon Alpha and Ribavirin Does Not Improve SVR in Patients with Genotypes 2/3 without Rapid Virological Response (OPTEX Trial): A Prospective, Randomized, Two-Arm, Multicentre Phase IV Clinical Trial. PLoS One. 2015 Jun 9;10(6):e0128069. doi: 10.1371/journal.pone.0128069. eCollection 2015. PMID 26057627
- See also: The network of competence for hepatitis (Hep-Net) will support the nation-wide research of viral hepatitis and will develop uniform diagnostic and therapeutic standards for five years. — http://www.kompetenznetz-hepatitis.de